CLINICAL TRIAL: NCT05002010
Title: Left Ventricular Hypertrophy Among Chronic Kidney Disease Patients in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Mohammed, Official title resident Doctor, Assiut University
Other Study IDs: LVH in CKD
Record Dates: First submitted 2021-07-24; First posted 2021-08-12 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Left Ventricular Hypertrophy; Chronic Kidney Diseases
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echo — Measure the Left ventricle (LV): IVS (interventricular septum), LVEDD(left ventricle end diastolic dimension ),LVESD((left ventricle end systolic dimension ), PWD(posterior wall dimension), LV systolic dysfunction and LV diastolic dysfunction.

SUMMARY:
Assess the prevalence and features of left ventricular hypertrophy in patients with chronic kidney disease (CKD) taking into account gender differences and stage of CKD.

To detect factors those predict LVH in CKD.

*to assess the right ventricle dysfunction in CKD .

DETAILED DESCRIPTION:
The number of patients with chronic kidney disease (CKD) is growing worldwide, while patients with impaired renal function are at high or very high risk for developing cardiovascular disease (CVD). Mortality due to CVD in patients with CKD is 1020 times higher than that in the general population, and the likelihood of developing cardiovascular complications (CVC) is several times higher than the risk of end-stage CKD{1} In CKD cardiovascular disease abnormalities are due to volume overload, hypertension, endothelia dysfunction, inflammation, uremic pericarditis cardiomyopathy, anemia, dyslipidemia and oxidativel stress{2} Left ventricular hypertrophy (LVH) is a key feature that allows you to get an accurate picture of systolic-diastolic lesions of the left heart in patients with CKD and therefore is one of the most important factors in the development of adverse CVC LVH is initially formed as an adaptive process aimed at maintaining normal heart function under conditions of myocardial overload by pressure or volume, but then acquires the character of pathological adaptation, becoming the structural basis of heart failure, myocardial ischemia and cardiac arrhythmias {3}. It was shown that the probability of LVH increases already with a moderate decrease in eGFR and increases further as CKD progresses, reaching a maximum in the terminal stage [4].

. in CKD LVH is associated with increased mortality and the risk of adverse outcomes, especially at the terminal stage of CKD{5-6}

ELIGIBILITY:
Inclusion Criteria:

- Patients with chronic renal disease (CKD) aged between 16 and 65 years will be included.

2- CKD are diagnosed based on criteria proposed by KDIGO (Kidney Disease: Improving Global Outcomes) in 2002

Exclusion Criteria:

* Patients with structural heart disease (congenital or valvular heart disease). Patients with primary hypertension. Patients with obstructive or restrictive lung disease.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Assess the prevalence and features of left ventricular hypertrophy in patients with chronic kidney disease (CKD) taking into account gender differences and stage of CKD.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Detecting the prevalence of LVH in CKD. | through study completion, an average of 1 year".
  The types of LVH in different stages of CKD. Risk factors of LVH in different stages of CKD

SECONDARY OUTCOMES:
The types of LVH in different stages of CKD. Risk factors of LVH in different stages of CKD | through study completion, an average of 1 year".

REFERENCES:
- [Background] Vallianou NG, Mitesh S, Gkogkou A, Geladari E. Chronic Kidney Disease and Cardiovascular Disease: Is there Any Relationship? Curr Cardiol Rev. 2019;15(1):55-63. doi: 10.2174/1573403X14666180711124825. PMID 29992892